CLINICAL TRIAL: NCT03945266
Title: Control Systems Engineering for Optimizing a Prenatal Weight Gain Intervention
Brief Title: Healthy Mom Zone: A Gestational Weight Gain Management Intervention
Acronym: HMZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Arizona State University (Other)
Responsible Party: Principal Investigator, Danielle Downs, Professor, Kinesiology and Obstetrics & Gyneocology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00003752; 5R01HL119245-05 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Overweight and Obesity; Physical Activity; Weight Change, Body; Eating Behavior
Keywords: gestational weight gain; pregnancy weight regulation; individually tailored intervention
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Body Weight Changes; Feeding Behavior; Gestational Weight Gain | interventions — Control Groups; Prenatal Care

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to an intervention or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive the allocated intervention to help manage gestational weight gain that includes education on weight regulation, healthy eating, physical activity, and goal setting.
  Interventions: Behavioral: Intervention group
- Control group (Active Comparator): Participants do not receive the allocated intervention but self-monitor their behaviors, complete study tasks and receive prenatal care as normal.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Intervention group — During the intervention, all participants will start out at the Baseline level. The baseline level will last 2 weeks and there will be an assessment to determine weight gain over those 2 weeks. If weight gain has succeeded the recommended amount, participants will be adapted up to a new level of intervention that includes education on GWG, healthy eating and physical activity. After every 4 weeks, an assessment will be performed and adaptations up will be made if necessary. Adaptations include addition of exercise sessions, healthy eating recipe demonstrations, and meal replacements. Participants will weigh themselves daily, wear an activity monitor, record their diet, and complete paper and online surveys.
  Arms: Intervention group
Behavioral: Control group — Participants will follow the same self-monitoring/assessment schedule but will not receive the GWG, healthy eating, and physical activity education or adaptations.
  Other Names: Prenatal care as usual
  Arms: Control group

SUMMARY:
The purpose is to establish feasibility of delivering an individually-tailored, behavioral intervention to manage gestational weight gain [GWG] that adapts to the unique needs and challenges of overweight/obese pregnant women [OW/OBPW] and will utilize control systems engineering to optimize this intervention; in other words, make this intervention manage GWG in OW/OBPW as effectively and efficiently as possible.

DETAILED DESCRIPTION:
The research proposed here will establish the dosage of components needed to impact GWG and develop an efficient (optimized) intervention to effectively manage GWG in OW/OBPW before a randomized controlled trial (RCT) can be implemented. The aims of the proposed research are: to establish feasibility of delivering an individually-tailored behavioral intervention for managing GWG in OW/OBPW. Two studies will be conducted to establish feasibility. Study 1 will examine viability of delivering dosages/sequencing of components (education, goal-setting, self-monitoring, HE/PA), GWG/HE/PA self-monitoring using e-health technology mechanisms, and data collection by delivering varied dosages to OW/OBPW over a brief, 4-week period followed by focus groups to evaluate user acceptability. The investigators will then make necessary revisions to the intervention. Study 2 will pilot test intervention delivery with decision rules for when/how to adapt dosages for an individual and randomization/retention/data collection procedures with treatment and control groups in a new cohort of OW/OBPW. Also, the investigators aim to use feasibility data collected from Aim 1 and control systems engineering to build a model that characterizes the effects of energy balance and planned/self-regulatory behaviors on GWG over time and use this model to develop an optimized intervention. The investigators will identify a dynamical model from feasibility data collected in Aim 1 that considers how changes in GWG responds to changes in energy intake, PA, and planned/self-regulatory behaviors. Model predictive control (a decision-making method from control systems engineering) will inform how the dosage adaptations are decided. The investigators will then identify a customized intervention plan for each woman based on her levels of energy intake, PA, planned/self-regulatory behaviors and the extent to which she is meeting GWG goals over pregnancy. This will lead to final program modifications and result in an individually-tailored, optimized intervention. The investigators will test the efficacy of this optimized intervention for managing GWG in OW/OBPW in a future RCT. This innovative research will develop an individually-tailored, optimized intervention that effectively and efficiently manages GWG in OW/OBPW and that will eventually be available to all pregnant women (via e-health technology) to improve the health of mothers and infants and impact the etiology of obesity and cardiovascular disease at a critical time in the life cycle.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Overweight or obese [body mass index range 24- >40 (if BMI (kg/m^2) is > 40, consultation with woman's health care provider (PCP/OBGYN) will be made to determine eligibility and ensure she does not have any contraindications to exercise) PI Danielle Downs will have communication with Dr. Hovick from MNPG to give information on the woman. The investigators also have a physician consent form (see Physician Patient Consent to Participate in documents) that the physician will complete as to whether the woman is eligible or not eligible to participate.
* Normal weight women with a BMI range of 18.0 to 23.9 can be enrolled in to the study as control participants (same measures of data collection, no opportunity for intervention).
* Ages 18-40 years [based on pilot data this group comprises >85% of the live births in Central Pennsylvania]
* 1st, 2nd or 3rd pregnancy 6-16 weeks gestation
* Able to read, understand, and speak English
* Residing in and around State College, PA
* 1st and 2nd time pregnant mothers [none or one other live or still born, biological children > 25 weeks gestation prior to this pregnancy; it may be conceivable that a woman has a blended family due to a mixed marriage and she will not be excluded if she is a parent to a guardian, foster child, or step child]
* Access to a computer or willingness to come onsite to complete study materials
* Infants born to participants who are 6-10 weeks old

Exclusion Criteria:

* Having more than one live or stillborn child > 25 weeks gestation; late-term pregnancy loss
* Diabetes at study entry [while future adaptations of this study will target women with diabetes, for the pilot study, they will be excluded to control for this confound]
* Contraindications to exercise in pregnancy [Hemodynamically significant heart disease, Restrictive lung disease, Incompetent cervix/cerclage, Persistent second [or third] trimester bleeding, Placenta previa after 26 weeks of gestation, Premature labor during the current pregnancy, Ruptured membranes, Preeclampsia/pregnancy-induced hypertension] per the ACOG guidelines [ACOG Committee on Obstetric Practice. [(2015, December). ACOG Committee opinion. Number 650: Physical Activity and Exercise During Pregnancy and the Postpartum Period. Obstetrics and Gynecology, 126,(6), 135-142].
* Having a body mass index less than 18 or over 40 (exclusion only if physician doesn't provide consent for BMI is over 40)
* Not planning to live in the area for the study duration
* Severe allergies or dietary restrictions that would preclude eating healthy foods
* Not able to read, understand, and/or speak English
* Cognitively impaired
* Currently smoking
* Infants not born to participants
* Infants younger than 6 weeks old

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle S Downs, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan per NIH guidelines per investigator user agreement and distribution agreement. Non-identified data, no hard-copy data can leave study site. Confidentiality agreements established.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Symons Downs D, Savage JS, Rivera DE, Smyth JM, Rolls BJ, Hohman EE, McNitt KM, Kunselman AR, Stetter C, Pauley AM, Leonard KS, Guo P. Individually Tailored, Adaptive Intervention to Manage Gestational Weight Gain: Protocol for a Randomized Controlled Trial in Women With Overweight and Obesity. JMIR Res Protoc. 2018 Jun 8;7(6):e150. doi: 10.2196/resprot.9220. PMID 29884603
- [Background] Guo P, Rivera DE, Pauley AM, Leonard KS, Savage JS, Downs DS. A "Model-on-Demand" Methodology For Energy Intake Estimation to Improve Gestational Weight Control Interventions. IFAC Pap OnLine. 2018;51(15):144-149. doi: 10.1016/j.ifacol.2018.09.105. Epub 2018 Oct 8. PMID 30480263
- [Background] Rauff EL, Downs DS. A Prospective Examination of Physical Activity Predictors in Pregnant Women with Normal Weight and Overweight/Obesity. Womens Health Issues. 2018 Nov-Dec;28(6):502-508. doi: 10.1016/j.whi.2018.09.003. Epub 2018 Oct 15. PMID 30337214
- [Background] Rauff EL, Downs DS. Mobile Health Technology in Prenatal Care: Understanding OBGYN Providers' Beliefs about Using Technology to Manage Gestational Weight Gain. J Technol Behav Sci. 2019 Mar;4(1):17-24. doi: 10.1007/s41347-018-0068-0. Epub 2018 Aug 15. PMID 30906851
- [Background] Pauley AM, Hohman E, Savage JS, Rivera DE, Guo P, Leonard KS, Symons Downs D. Gestational Weight Gain Intervention Impacts Determinants of Healthy Eating and Exercise in Overweight/Obese Pregnant Women. J Obes. 2018 Oct 1;2018:6469170. doi: 10.1155/2018/6469170. eCollection 2018. PMID 30364005
- [Background] Guo P, Rivera DE, Savage JS, Hohman EE, Pauley AM, Leonard KS, Downs DS. System Identification Approaches For Energy Intake Estimation: Enhancing Interventions For Managing Gestational Weight Gain. IEEE Trans Control Syst Technol. 2020 Jan;28(1):63-78. doi: 10.1109/TCST.2018.2871871. Epub 2018 Oct 12. PMID 31903018
- [Background] Freigoun MT, Rivera DE, Guo P, Hohman EE, Gernand AD, Downs DS, Savage JS. A Dynamical Systems Model of Intrauterine Fetal Growth. Math Comput Model Dyn Syst. 2018;24(6):661-687. doi: 10.1080/13873954.2018.1524387. Epub 2018 Oct 7. PMID 30498392
- [Background] Guo P, Rivera DE, Savage JS, Downs DS. State Estimation Under Correlated Partial Measurement Losses: Implications for Weight Control Interventions. IFAC Pap OnLine. 2017 Jul;50(1):13532-13537. doi: 10.1016/j.ifacol.2017.08.2347. Epub 2017 Oct 18. PMID 29242854
- [Background] Downs DS. Obesity in Special Populations: Pregnancy. Prim Care. 2016 Mar;43(1):109-20, ix. doi: 10.1016/j.pop.2015.09.003. Epub 2016 Jan 12. PMID 26896204
- [Background] Devlin CA, Huberty J, Downs DS. Influences of prior miscarriage and weight status on perinatal psychological well-being, exercise motivation and behavior. Midwifery. 2016 Dec;43:29-36. doi: 10.1016/j.midw.2016.10.010. Epub 2016 Oct 29. PMID 27838526
- [Background] Guo P, Rivera DE, Downs DS, Savage JS. Semi-physical Identification and State Estimation of Energy Intake for Interventions to Manage Gestational Weight Gain. Proc Am Control Conf. 2016 Jul;2016:1271-1276. doi: 10.1109/ACC.2016.7525092. Epub 2016 Aug 1. PMID 27570366
- [Background] Downs DS, Devlin CA, Rhodes RE. The Power of Believing: Salient Belief Predictors of Exercise Behavior in Normal Weight, Overweight, and Obese Pregnant Women. J Phys Act Health. 2015 Aug;12(8):1168-76. doi: 10.1123/jpah.2014-0262. Epub 2014 Nov 19. PMID 25409425
- [Background] Savage JS, Downs DS, Dong Y, Rivera DE. Control systems engineering for optimizing a prenatal weight gain intervention to regulate infant birth weight. Am J Public Health. 2014 Jul;104(7):1247-54. doi: 10.2105/AJPH.2014.301959. Epub 2014 May 15. PMID 24832411
- [Background] Dong Y, Deshpande S, Rivera DE, Downs DS, Savage JS. Hybrid Model Predictive Control for Sequential Decision Policies in Adaptive Behavioral Interventions. Proc Am Control Conf. 2014 Jun;2014:4198-4203. doi: 10.1109/ACC.2014.6859462. PMID 25635157
- [Background] Downs DS, Savage JS, Rauff EL. Falling Short of Guidelines? Nutrition and Weight Gain Knowledge in Pregnancy. J Womens Health Care. 2014;3:1000184. doi: 10.4172/2167-0420.1000184. PMID 25599012
- [Background] Dong Y, Rivera DE, Downs DS, Savage JS, Thomas DM, Collins LM. Hybrid Model Predictive Control for Optimizing Gestational Weight Gain Behavioral Interventions. Proc Am Control Conf. 2013:1970-1975. doi: 10.1109/acc.2013.6580124. PMID 24336314
- [Background] Dong Y, Rivera DE, Thomas DM, Navarro-Barrientos JE, Downs DS, Savage JS, Collins LM. A Dynamical Systems Model for Improving Gestational Weight Gain Behavioral Interventions. Proc Am Control Conf. 2012:4059-4064. doi: 10.1109/acc.2012.6315424. PMID 24309837
- [Background] McNitt KM, Hohman EE, Rivera DE, Guo P, Pauley AM, Gernand AD, Symons Downs D, Savage JS. Underreporting of Energy Intake Increases over Pregnancy: An Intensive Longitudinal Study of Women with Overweight and Obesity. Nutrients. 2022 Jun 1;14(11):2326. doi: 10.3390/nu14112326. PMID 35684126
- [Background] Rosinger AY, Bethancourt HJ, Pauley AM, Latona C, John J, Kelyman A, Leonard KS, Hohman EE, McNitt K, Gernand AD, Downs DS, Savage JS. Variation in urine osmolality throughout pregnancy: a longitudinal, randomized-control trial among women with overweight and obesity. Eur J Nutr. 2022 Feb;61(1):127-140. doi: 10.1007/s00394-021-02616-x. Epub 2021 Jul 3. PMID 34218315
- [Background] Guo P, Rivera DE, Dong Y, Deshpande S, Savage JS, Hohman EE, Pauley AM, Leonard KS, Downs DS. Optimizing Behavioral Interventions to Regulate Gestational Weight Gain With Sequential Decision Policies Using Hybrid Model Predictive Control. Comput Chem Eng. 2022 Apr;160:107721. doi: 10.1016/j.compchemeng.2022.107721. Epub 2022 Feb 8. PMID 35342207
- [Background] Leonard KS, Pauley AM, Hohman EE, Guo P, Rivera DE, Savage JS, Buman MP, Symons Downs D. Identifying ActiGraph non-wear time in pregnant women with overweight or obesity. J Sci Med Sport. 2020 Dec;23(12):1197-1201. doi: 10.1016/j.jsams.2020.08.003. Epub 2020 Aug 11. PMID 32859522
- [Background] Ranghetti L, Rivera DE, Guo P, Visioli A, Savage JS, Symons Downs D. A control-based observer approach for estimating energy intake during pregnancy. Int J Robust Nonlinear Control. 2023 Jun;33(9):5105-5127. doi: 10.1002/rnc.6019. Epub 2022 Jan 30. PMID 37193543
- [Result] Savage JS, Hohman EE, McNitt KM, Pauley AM, Leonard KS, Turner T, Pauli JM, Gernand AD, Rivera DE, Symons Downs D. Uncontrolled Eating during Pregnancy Predicts Fetal Growth: The Healthy Mom Zone Trial. Nutrients. 2019 Apr 21;11(4):899. doi: 10.3390/nu11040899. PMID 31010102
- [Result] Downs DS, Savage JS, Rivera DE, Pauley AM, Leonard KS, Hohman EE, Guo P, McNitt KM, Stetter C, Kunselman A. Adaptive, behavioral intervention impact on weight gain, physical activity, energy intake, and motivational determinants: results of a feasibility trial in pregnant women with overweight/obesity. J Behav Med. 2021 Oct;44(5):605-621. doi: 10.1007/s10865-021-00227-9. Epub 2021 May 5. PMID 33954853
- [Result] Leonard KS, Symons Downs D. Low prenatal resting energy expenditure and high energy intake predict high gestational weight gain in pregnant women with overweight/obesity. Obes Res Clin Pract. 2022 Jul-Aug;16(4):281-287. doi: 10.1016/j.orcp.2022.07.003. Epub 2022 Jul 13. PMID 35840506
- [Result] Pauley AM, Hohman EE, Leonard KS, Guo P, McNitt KM, Rivera DE, Savage JS, Downs DS. Short Nighttime Sleep Duration and High Number of Nighttime Awakenings Explain Increases in Gestational Weight Gain and Decreases in Physical Activity but Not Energy Intake among Pregnant Women with Overweight/Obesity. Clocks Sleep. 2020 Nov 14;2(4):487-501. doi: 10.3390/clockssleep2040036. PMID 33202691
- [Derived] Hohman EE, Smyth JM, McNitt KM, Pauley AM, Symons Downs D, Savage JS. Urinary cortisol is lower in pregnant women with higher pre-pregnancy BMI. Front Endocrinol (Lausanne). 2023 Jan 11;13:1014574. doi: 10.3389/fendo.2022.1014574. eCollection 2022. PMID 36714602
- See also: Youtube video describing the intervention — https://youtu.be/7Zqmgw_Cuss?list=PLXtTiUbk7YSArO9xX3wHp0YO2IPt3qKR0

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 15 | 16
Completed | 13 | 14
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Miscarriage | 0 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (3.7) | 29.6 (4.5) | 29.6 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
Pre-pregnancy BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.4 (7.6) | 32.7 (7.0) | 32.6 (7.2)
Pre-pregnancy Weight [Mean (Standard Deviation); unit: kilograms] | 86.4 (20.0) | 91.2 (22.4) | 88.9 (21.0)
Weight at Study Enrollment [Mean (Standard Deviation); unit: kilograms] | 87.2 (19.8) | 92.4 (21.0) | 89.9 (20.2)
Gestational Age [Mean (Standard Deviation); unit: weeks] | 10.3 (1.6) | 10.1 (1.7) | 10.2 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Gestational Weight Change
Description: Gestational weight change will be measured daily at home using the FitBit Aria Wi-Fi Smart Scale (www.fitbit.com; weights will be wirelessly uploaded to online program). Gestational weight change will be standardized: target weight gain will be determined for each woman based on BMI (kg/m^2) status (OW = 15-25 lb, OB = 11-20 lb). For the criterion measure to determine when to adapt the intervention, weight gain will be calculated to determine if a woman is gaining < her goal (-), at the exact amount of her goal (0), or > her goal (+). Pre-pregnancy weight and gestational weight change from the first prenatal visit to the last pre-delivery weight will also be obtained from clinical records. Overweight/obese pregnant women (OW/OBPW) often exceed the GWG guidelines, managing weight gain in this population is critical. Participants weigh themselves daily using a WiFi connected scale. Outcome measure reported at mean change from pre- to post-intervention.
Time Frame: Daily data was collected starting at baseline (pre-intervention), through study completion Month 6 (post-intervention). Also measured daily for one week at 6-weeks postpartum. Outcome measure reported at mean change from pre- to post-intervention.
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
kilograms | 6.9 [3.8 to 10.0] | 8.8 [5.1 to 12.3]

2. Secondary Outcome: Theory of Planned Behavior (Motivational Determinants of Healthy Eating)
Description: The Theory of Planned Behavior will inform our dynamical model in order to create individualized interventions for OW/OBPW. Beliefs: These items were developed to assess Theory of Planned Behavior (TPB) behavioral, control, and normative beliefs. Main Constructs: The Theory of Planned Behavior (TPB) Healthy Eating Main Constructs measure is a 38-item measure developed to assess the main constructs of the TPB (i.e., attitude, subjective norm (SN), perceived behavioral control (PBC), intention) as they relate to healthy eating behavior. Scoring for the TPB is the sum of each subscale. Attitude and Limit Attitude range of scores: 7-49 - higher score means greater/more positive attitude; SN and Limit SN range: 3-21 - higher score greater/more positive subjective norm; PBC and Limit PBC range: 3-21 - higher score greater/more positive PBC; Intention range: 6-42 - higher score greater/more positive intention. Results reported reflect mean changes from pre-intervention to post-intervention.
Time Frame: Data was collected each month starting at baseline (pre-intervention), through study completion at Month 6 (post-intervention). Pre-intervention, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, post-intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
score on a scale
  Attitude | -1.8 [-4.2 to 0.6] | -2.5 [-4.8 to -0.2]
  Subjective Norm | 0.0 [-1.4 to 1.4] | -1.4 [-2.7 to -0.1]
  Perceived Behavioral Control | -0.8 [-2.1 to 0.4] | -0.3 [-1.5 to 0.9]
  Intention | -2.1 [-4.8 to 0.7] | -3.2 [-5.8 to -0.7]
  Limit Unhealthy Eating Attitude | -0.2 [-3.4 to 2.9] | -0.9 [-3.9 to 2.0]
  Limit Unhealthy Eating Subjective Norm | 0.0 [-2.7 to 0.6] | -0.9 [-2.6 to 0.8]
  Limit Unhealthy Eating Perceived Behavioral Control | 0.0 [-1.6 to 1.7] | -0.8 [-2.4 to 0.8]
  Limit Unhealthy Eating Intention | -0.6 [-3.9 to 2.6] | -2.9 [-6.0 to 0.3]

3. Secondary Outcome: Theory of Planned Behavior (Motivational Determinants of Physical Activity)
Description: The Theory of Planned Behavior will inform our dynamical model in order to create individualized interventions for OW/OBPW. Beliefs: These items were developed to assess Theory of Planned Behavior (TPB) behavioral, control, and normative beliefs. Main Constructs: The Theory of Planned Behavior (TPB) Healthy Eating Main Constructs measure is a 38-item measure developed to assess the main constructs of the TPB (i.e., attitude, subjective norm (SN), perceived behavioral control (PBC), intention) as they relate to healthy eating behavior. Scoring for the TPB is the sum of each subscale. Attitude range of scores: 7-49 - higher score means greater/more positive attitude; SN range: 3-21 - higher score greater/more positive subjective norm; PBC range: 3-21 - higher score greater/more positive PBC; Intention range: 6-42 - higher score greater/more positive intention. Results reported reflect mean changes from pre-intervention to post-intervention.
Time Frame: Data was collected each month starting at baseline (pre-intervention), through study completion at post-intervention - Pre-intervention, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, post-intervention.
Measure: Mean (95% Confidence Interval); unit: change score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
change score on a scale
  Physical Activity Attitude | -2.9 [-8.2 to 2.5] | -1.1 [-6.2 to 3.9]
  Physical Activity Subjective Norm | -0.2 [-3.0 to 2.5] | 0.3 [-2.3 to 2.9]
  Physical Activity Perceived Behavioral Control | -0.7 [-3.0 to 1.5] | 1.5 [-0.7 to 3.7]
  Physical Activity Intention | 1.8 [-1.2 to 4.7] | -1.9 [-4.9 to 1.0]

4. Secondary Outcome: Self-regulation of Healthy Eating
Description: Self-regulation of HE will be measured in order to inform our dynamical model and to how well OW/OBPW are at regulating their energy intake and expenditure and how it impacts their GWG.
  These items were taken from Ryan Rhodes items for self-regulation of PA and adapted for HE behaviors. Ryan has indicated that these items work really well as an index for HE self-regulation because these behaviors are naturally inter-connected but to look at specific self-regulatory behaviors: self-monitoring, goal-setting, action planning, coping planning, scheduling, affective There are also 2 sets of 8 questions-first 8 examine prospective behaviors while the second set assesses retrospective behaviors.
  Retrospective scores range from 11-55 and Prospective scores range from 11-55. Total scores range from 22-110. A higher score indicates higher levels of HE self-regulation. Results are mean difference of pre- and post-intervention week.
Time Frame: Data was collected bi-weekly starting at baseline (pre-intervention), through study completion at Month 6 (post-intervention). Pre-intervention week, week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, and post-intervention week.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
score on a scale
  Healthy Eating Prospective Self-Regulation | -3.3 [-6.9 to 0.4] | -3.5 [-7.1 to 0.1]
  Healthy Eating Retrospective Self-Regulation | 1.6 [-3.0 to 6.1] | 4.5 [-0.1 to 9.0]

5. Secondary Outcome: Self-regulation of Physical Activity
Description: Self-regulation of PA will be measured in order to inform our dynamical model and to how well OW/OBPW are at regulating their energy intake and expenditure and how it impacts their GWG. These items are taken from Ryan Rhodes. Ryan has indicated that these items work really well as an index because these behaviors are naturally inter-connected but to look at specific self-regulatory behaviors: Item #1: self-monitoring, Item #2: goal-setting, Item # 3: action planning, Item #4: coping planning, Item #5: scheduling, Item #6, 7, 8, 9: cuing, Items 10 & 11: affective. There are also 2 sets of 8 questions-first 8 examine prospective behaviors while the second set assesses retrospective behaviors. Retrospective scores range from 11-55 and Prospective scores range from 11-55. Total scores for overall self-regulation range from 22-110. A higher score indicates higher levels of PA self-regulation. Results reported reflect mean changes from pre to post-intervention week.
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
score on a scale
  Physical Activity Prospective Self-Regulation | -1.3 [-5.0 to 2.3] | -4.9 [-8.4 to -1.4]
  Physical Activity Retrospective Self-Regulation | 5.6 [1.2 to 10.1] | 0.3 [-4.0 to 4.7]

6. Secondary Outcome: Objective Activity Monitor UP Jawbone
Description: Women will be wearing the UP Jawbone for the entire six week intervention. UP will track how the participants sleep, move and eat. Women will be wearing the UP Jawbone in counterbalance with the Actigraph wGt3X-BTI. The specific outcome measure used from the activity monitor is calories (kcals) burned during physical activity/exercise. Outcome measure reported at mean change from pre- to post-intervention.
Time Frame: Daily data was collected starting at pre-intervention, through study completion post-intervention. Daily for a total of 6 months. Outcome measure reported at mean change from pre- to post-intervention.
Measure: Mean (95% Confidence Interval); unit: calories per day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
calories per day | 34.9 [-245.6 to 315.4] | -78.9 [-273.5 to 115.7]

7. Secondary Outcome: Energy Intake
Description: Estimated energy intake (kcals) from physical activity (kcals) and weight (GWG). Outcome measure reported as mean change of energy intake calories from pre to post-intervention.
Time Frame: Daily energy intake was estimated starting at pre-intervention through post-intervention. Each day for 6 months. Outcome measure reported as mean change of energy intake calories from pre to post-intervention.
Measure: Mean (95% Confidence Interval); unit: calories per day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
calories per day | 410.2 [32.4 to 787.9] | 1134.8 [697.3 to 1572.3]

8. Secondary Outcome: MyFitnessPal
Description: MyFitness Pal: Web-based and smartphone app dietary intake tracker. Women tracked their diets every day for 6 months and every day for one week at their 6 week postpartum period. Energy intake or calories (kcal) consumed each day were measured. Outcome measure reported as mean change of energy intake calories from pre to post-intervention.
Time Frame: Data was collected 3 days a week, each week from pre-intervention through post-intervention. A total of 72 days over 6 months. Outcome measure reported as mean change of energy intake calories from pre-intervention week to post-intervention week.
Measure: Mean (Standard Deviation); unit: calories per day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 9 | 10
calories per day | 1541.5 (372.9) | 1402.2 (413.3)

9. Secondary Outcome: Three Factor Eating Questionnaire
Description: The Three Factor Eating Questionnaire is a 51-item questionnaire to measure three dimensions of human eating behavior: 1) dietary restraint, or cognitive control of eating behavior, 2) dietary disinhibition, or disinhibition of cognitive control of eating, and 3) susceptibility to hunger. The investigators are only using 18 items of the revised TFEQ. These items are known as TFEQ-R18 as reported in (de Lauzon et al., 2004). The TFEQ is examined by subscale scores and not by a total score. Subscale scores for the cognitive restraint scale range from 3-12; higher scores indicate higher levels of cognitive restraint of eating. Uncontrolled eating scale range from 9-36; higher scores indicate higher levels of uncontrolled eating behaviors. Emotional eating scale range from 6-24; higher scores indicate higher levels of emotional eating behaviors. Outcome measure results are reported as the score during the post-intervention week.
Time Frame: Data was collected monthly starting at pre-intervention, through post-intervention - Pre-intervention, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 11 | 12
score on a scale
  Cognitive Restraint | 7.3 (1.7) | 7.5 (1.9)
  Emotional Eating | 11.2 (4.5) | 12.3 (3.98)
  Uncontrolled Eating | 19.1 (6.8) | 17.0 (3.2)

10. Secondary Outcome: Leisure Time Exercise Questionnaire
Description: The Leisure-Time Exercise Questionnaire (LTEQ) is a 3 item questionnaire to measure the amount and intensity of exercise a person engages in during a one week period. Reported scores are multiplied by 15 to get total min/week for each type and then adding those values together to total min of weekly exercise. Higher scores reflect more minutes of physical activity. Results reported reflect mean changes from pre- to post-intervention.
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 10 | 10
minutes/week | 315 (399.0) | 184.5 (272.2)

11. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: Pittsburgh Sleep Quality Index: The Pittsburgh Sleep Quality Index (PSQI) is an 18-item measure developed by Smyth (2003) to measure the quality and patterns of sleep in older adults. It differentiates "poor" from "good" sleep by measuring seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction over the last month. Scores can range from 0-21. An overall sleep quality score greater than or equal to 5 reflects poor sleep quality. The outcome reported is overall sleep quality. Results reported reflect mean at post-intervention.
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 9 | 12
score on a scale | 7.0 (3.6) | 6.1 (2.9)

12. Secondary Outcome: Sleep Behaviors (Activity Monitor) - Nighttime Sleep Duration
Description: UP Jawbone activity monitor: women wear the monitor during the night and measures sleep duration. This outcome reports mean nighttime sleep duration over the entire study duration.
Time Frame: Data was collected each day starting at pre-intervention, through post-intervention - a total of 6 months of daily data collection.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
minutes | 414.5 (45.2) | 451.3 (74.2)

13. Secondary Outcome: Fetal Measure: Ultrasounds [Fetal Growth]
Description: Ultrasounds are conducted each month to measure fetal growth. Ultrasounds were completed for fetal growth measures as well to ensure adequate growth for those in the study. If there were any flags for growth restriction concerns, participant's physicians were alerted. These ultrasounds were used as safety checks and to ensure proper fetal growth. No group analyses were conducted nor were there any comparisons between groups. Data reported is the sum of all flagged ultrasounds over the study duration.
Time Frame: Each month - Month 1, Month 2, Month 3, Month 4, Month 5, and Month 6. Data reported is the sum of all flagged ultrasounds over the study duration.
Measure: Number; unit: ultrasounds
Groups:
- Intervention: Participants receive the allocated intervention to help manage gestational weight gain that includes education on weight regulation, healthy eating, physical activity, and goal setting.
  Intervention group: During the intervention, all participants will start out at the Baseline level. The baseline level will last 2 weeks and there will be an assessment to determine weight gain over those 2 weeks. If weight gain has succeeded the recommended amount, participants will be adapted up to a new level of intervention that includes education on GWG, healthy eating and physical activity. After every 4 weeks, an assessment will be performed and adaptations up will be made if necessary. Adaptations include addition of exercise sessions, healthy eating recipe demonstrations, and meal replacements. Participants will weigh themselves daily, wear an activity monitor, record their diet, and complete paper and online surveys.
- Control: Participants do not receive the allocated intervention but self-monitor their behaviors, complete study tasks and receive prenatal care as normal.
  Control group: Participants will follow the same self-monitoring/assessment schedule but will not receive the GWG, healthy eating, and physical activity education or adaptations.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 14
ultrasounds | 8 | 0

14. Secondary Outcome: Infant Birthweight
Description: The infant's birth weight will be obtained through medical records or self-report from mother.
Time Frame: Assessed at time of birth - data abstracted at 6-week postpartum session.
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Intervention: Birth weights were extracted for each intervention participant's infant through electronic health record data.
- Control: Birth weights were extracted for each control participant's infant through electronic health record data.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 13
grams | 3379.7 (628.5) | 3266.4 (672.6)

15. Secondary Outcome: Infant Length
Description: The infant's birth length will be obtained through medical records or self-report from mother
Time Frame: Assessed at time of birth - data abstracted at 6-week postpartum session.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 7 | 7
centimeters | 43.9 (1.9) | 52.5 (2.6)

16. Secondary Outcome: Resting Metabolic Rate
Description: The Breezing Device: An indirect calorimetry analyzer that measures the rate of oxygen consumption and carbon dioxide production and determines how much energy the body is burning due to the metabolism of nutrients (named Resting Energy Expenditure, REE), and the type of nutrients the body uses to produce energy (Energy source = respiratory quotient, RQ). Developed at Arizona State University. The Breezing is a cellphone-size, battery operated, portable technology that syncs with smartphones. This tracker takes a traditional laboratory-based measurement and makes it faster, more affordable and mobile. Breezing has a 99.8% correlation with the gold standard method, Douglas Bag. Outcome measure is reported as an average over the entire study period.
Time Frame: Data was collected weekly from pre-intervention to post-intervention - Pre-intervention, week 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 ,15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, post-intervention.
Measure: Mean (Standard Deviation); unit: kcals/day
Arm/Group | Intervention | Control Group
Number analyzed (Participants) | 8 | 12
kcals/day | 1861.12 (297.46) | 1867.10 (324.35)

17. Secondary Outcome: Body Area Satisfaction Scale
Description: The Body Area Satisfaction Scale (BASS) measure is a 9-item subscale originating from the Multidimensional Body-Self Relations Questionnaire (MBSRQ), which is a 69-item self-report inventory for the assessment of self-attitudinal aspects of the construct of body-image. The BASS assesses one's personal satisfaction with body parts such as arms, legs, and face in which participants rate their degree of body satisfaction with each specified body party from 1 (very dissatisfied) to 5 (very satisfied). The first 8 of the 9 items are added together for a total score. Scores range from 8-40. A higher score indicates higher body satisfaction. Outcome measure is reported as the score at post-intervention.
Time Frame: Data was collected monthly starting at pre-intervention, through study post-intervention - Pre-intervention, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and post-intervention. Outcome measure is reported as the score at post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 11 | 12
score on a scale | 25.2 (3.6) | 23.5 (4.6)

18. Secondary Outcome: Center for Epidemiological Studies Depression Scale
Description: Center for Epidemiological Studies Depression Scale (CESD): Measures current levels of depressive symptomology. A cut off score of 16 is used to determine case status (depressed versus not depressed). A higher score (above 16) represents depressive symptomology. A total CES-D score can be calculated [Total CES-D Score = sum (items 1-20)]. Scores range from 0-60. Outcome reported is the mean scores at the post-intervention time period.
Time Frame: Data was collected monthly starting at pre-intervention, through study post-intervention - Pre-intervention, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and post-intervention. Results are the mean scores at the post-intervention time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 14
score on a scale | 10.6 (8.0) | 8.1 (5.1)

19. Secondary Outcome: State-Trait Anxiety Inventory
Description: The State-Trait Anxiety Inventory (STAI) is a 20-item questionnaire to measure state and trait anxiety. The State version of the STAI is being used for the current study. This scale consists of twenty items that evaluate how respondents feel "right now, at this moment." In responding to the STAI State-Anxiety scale, participants choose the response statement that best describes the intensity of their feelings: (1) not at all; (2) somewhat; (3) moderately so; (4) very much so. The state version of the STAI can also be used to evaluate how someone felt at a particular time in the recent past and how they anticipated to feel either in a specific situation that is likely to be encountered in the future or in a variety of hypothetical situations. Scores can range: 20-80. A total score is used to determine anxiety. A higher score indicates higher anxiety. Outcome reported is the mean scores at the post-intervention time period.
Time Frame: Data was collected monthly starting at pre-intervention through post-intervention: Pre-intervention, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, and Post-intervention. Results reported reflect mean scores at the post-intervention time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 11 | 12
score on a scale | 36.1 (13.3) | 29.0 (9.7)

20. Secondary Outcome: Perceived Stress Scale
Description: The Perceived Stress Scale (PSS) is a 10-item scale developed by Cohen (1988) that measures the degree to which situations in one's life are appraised as stressful. The PSS was designed for use with community samples with at least a junior high-school education. The 14 items are easy to understand and the response alternatives (never, almost never, neutral, sometimes, fairly often, very often) are simple to grasp. The questions are quite general in nature and hence relatively free of content specific to any sub-population group. Scores range from 0-40. A higher score indicates higher levels of perceived stress.
Time Frame: Assessed weekly at pre-intervention week, week 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, and post-intervention. Post-intervention mean scores reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 14
score on a scale | 25 (8.6) | 23.2 (7.2)

21. Secondary Outcome: Sleep Behaviors (Activity Monitor) - Nighttime Awakenings
Description: UP Jawbone activity monitor: women wear the monitor during the night. The monitor measures number of awakenings. This outcome reports mean nighttime awakenings per night over the entire study duration (pre- to post-intervention).
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: nighttime awakenings
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 14
nighttime awakenings | 1.8 (.7) | 1.7 (.8)

ADVERSE EVENTS:
Time Frame: Tracking of adverse events was done over a 6 month period.
Description: Adverse events were tracked/collected if any woman experienced any obstetric issues with the physical activity sessions or healthy eating demonstrations. Our protocol stated that ALL physical activity sessions and healthy eating demonstrations were performed and monitored by a certified prenatal exercise specialist or a registered dietician and all sessions were monitored by a Penn State employed nurse and a member of the study team. Any events were immediately reported to the PI and the IRB.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 8/15 | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=15) | Control Group (N=16)
Fetal Growth and Abnormalities (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 0 (0) — Ultrasounds were performed on a monthly basis. Study team physicians review each ultrasound for any issues. If flagged, participant's physicians are notified and provided additional medical screening/care, if necessary. All non-study related.
Depressive Symptoms (Psychiatric disorders) | 1 (1) | 3 (3) — All women complete the CESD. If scores >16, women are provided a consult with a study nurse practitioner. All participants are provided with local psychological care resources.
Gestational Diabetes (Metabolism and nutrition disorders) | 1 (1) | 3 (3) — Participants self-report GDM diagnoses during study participation or GDM diagnoses determined through electronic health record extraction. Participants are still able to participate but study staff are in contact with physicians.
Maternal Blood Draw and Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) — Pre and post blood draws are monitored for any bruising, blood flow, or anemia concerns. Follow-ups with physicians are required for each event.

LIMITATIONS AND CAVEATS:
We were not adequately powered to detect significant effects on secondary outcomes due to the feasibility study design.

Our sample was largely homogenous (Caucasian, middle income, well educated).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT03945266/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03945266/ICF_001.pdf